CLINICAL TRIAL: NCT06414044
Title: STudio Osservazionale Sull'Efficacia, Sicurezza e tollerabilità di Atogepant in Pazienti Real Life Affetti da Emicrania in Italia (Studio STAR)
Brief Title: Italian Real-life obServational Study on the effecTiveness, sAfety and Tolerability of Atogepant in Migraine Patients
Acronym: STAR
Status: Active, not recruiting | Type: Observational
Sponsor: University of Florence (Other)
Collaborators: Fondazione Policlinico Universitario Campus Bio-Medico (Other); IRCCS National Neurological Institute "C. Mondino" Foundation (Other); Società Italiana per lo Studio delle Cefalee (Other); Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other); Università degli Studi dell'Aquila (Other); University of Roma La Sapienza (Other); Azienda Ospedaliero Universitaria Policlinico Modena (Other); Euganea Health Unit, Padua, Italy (Unknown); Azienda Ospedaliero-Universitaria di Parma (Other); Azienda Ospedaliera S. Maria della Misericordia (Other); A.O.U. Città della Salute e della Scienza (Other); Cliniche Humanitas Gavazzeni (Other); University of Campania Luigi Vanvitelli (Other); Ospedale Santo Stefano (Other); Azienda Policlinico Umberto I (Other); Auxologico San Luca (Other); Asst Degli Spedali Civili Di Brescia (Other)
Responsible Party: Principal Investigator, Luigi Francesco Iannone, Researcher at the Headache Center and Clinical Pharmacology Unit and at the Department of Health Sciences, University of Florence, Principal Investigator, University of Florence
Other Study IDs: RICe_4
Record Dates: First submitted 2024-05-10; First posted 2024-05-14 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Migraine; Migraine With Aura; Migraine Without Aura; Chronic Migraine
Keywords: Headache; Medication overuse headache; Pain; Migraine prevention; Gepant
MeSH Terms: conditions — Migraine Disorders; Migraine with Aura; Migraine without Aura; Headache; Headache Disorders, Secondary; Pain | interventions — atogepant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Episodic migraine: Patients affected by migraine with an episodic pattern (< 15 monthly migraine days) with or without aura according to ICHD-III criteria.
  Interventions: Drug: Atogepant 60 mg
- Chronic migraine: Patients affected by chronic migraine (> 15 monthly headache days with at least 8 days with migraine features) according to ICHD-III criteria.
  Interventions: Drug: Atogepant 60 mg

INTERVENTIONS:
Drug: Atogepant 60 mg — Patients using atogepant 60 mg tablet daily as migraine prevention

SUMMARY:
The purpose of this prospective and multicentric study is to evaluate the effectiveness and tolerability of atogepant as preventive migraine treatment in a cohort of episodic or chronic migraine patients.

DETAILED DESCRIPTION:
Atogepant is a small molecule calcitonin gene- related peptide (CGRP) receptor antagonist, part of the gepants family. It is a second generation gepant, currently approved for the preventive treatment of episodic and chronic migraine.

Previously randomized, placebo-controlled phase 2/3 trials demonstrated its effectiveness and tolerability in the preventive setting for patients with episodic and chronic migraine, associated with a good tolerability profile.

The most commonly reported adverse events were upper respiratory tract infections, urinary infections, nausea and constipation.

In this prospective multicentric study the investigators aim to evaluate atogepant effectiveness and tolerability as preventive migraine treatment in a real-world setting. Subjects who meet the inclusion criteria will be enrolled and will participate in the study. Baseline demographic and clinical data will be collected at the baseline.

patients will take atogepant 60 mg daily for at least 12 weeks up to two years, according to effectiveness, tolerability and eventual approval of reimbursability criteria.

Data will be collected at baseline and every three months for two years. Subjects will be asked to keep a headache diary to collect monthly headache and migraine days, migraine severity, associated symptoms and drug consumption. Questionnaires will be collected every three months.

Data collection will focus on: i) demographic data, ii) migraine history, iii) pain intensity, iv) presence and evolution of migraine associated symptoms and aura, v) migraine associated disability, vi) tolerability and eventual treatment- emergent adverse events, vii) treatment persistence. The online database REDCap will be used for data collection.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraine without aura, migraine with aura, or chronic migraine according to the 3rd edition of the International Classification of Headache Disorder (ICHD-III);
* At least 3 monthly migraine days;
* Good compliance to study procedures;
* Availability of headache diary at least of the preceding months before enrollment.

Exclusion Criteria:

* Subjects with contraindications for use of gepants;
* Concomitant diagnosis of medical diseases and/or comorbidities that, in the Investigator's opinion might interfere with study assessments;
* medical comorbidities that could interfere with study results;
* Pregnancy and breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multicentric study on patients attending the outpatient clinic of Italian Headache centres who meet criteria for atogepant use for migraine preventive treatment.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2024-05-09 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Changes in migraine frequency after three months of treatment | Baseline (T0) - 3 months of treatment with atogepant (T3)
  Changes in monthly migraine days after three months of treatment with atogepant compared to baseline (continuous variable)
50% Response after three months of treatment | Baseline (T0) - 3 months of treatment with atogepant (T3)
  Percentage of 50% Responders (namely patients who presented a reduction of MMDs >/ = 50% compared to baseline) after three months of treatment with atogepant (continuous variable)

SECONDARY OUTCOMES:
Changes in migraine frequency across twelve months of atogepant treatment | Baseline (T0) - 6 months (T6) - 12 months (T12) of treatment with atogepant
  Changes in monthly migraine days after six and twelve months of treatment with atogepant compared to baseline (continuous variable)
Percentage of 50% Responders (namely patients who presented a reduction of MMDs >/ = 50% compared to baseline) across twelve months of treatment with atogepant | Baseline (T0) - 6 months (T6) - 12 months (T12) of treatment with atogepant
  Percentage of 50% Responders (namely patients who presented a reduction of MMDs >/ = 50% compared to baseline) after six and twelve months of treatment with atogepant (continuous variable)
Evaluation of any adverse event (qualitative) | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with atogepant
  Type of any adverse events in patients receiving atogepant during the observation period (categorical variable)
Evaluation of any adverse event (quantitative) | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with atogepant
  Percentage of reported adverse events in patients receiving atogepant assessed quarterly during the observation period (continuous variable)
Evaluation of serious adverse event | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with atogepant
  Percentage of serious adverse events (namely those resulting in death, is life-threatening, requires hospitalisation or prolongation of existing hospitalisation, results in persistent or significant disability or incapacity, or is a birth defect) in patients receiving atogepant during the observation period (continuous variable)
Evaluation of adverse event leading to treatment discontinuation | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with atogepant
  Percentage of adverse events leading to treatment discontinuation in patients receiving atogepant during the observation period (continuous variable)
Consistency of treatment response | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with atogepant
  Percentage of patients with a stable 50% response across twelve months of atogepant treatment (continuous variable)
Changes in migraine disability (MIDAS) | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with atogepant
  Changes in MIgraine Disability ASsement questionnaire across treatment (continuous variable, 0-270 scale, higher scores indicate higher disability: 0-5, little/no disability; 6-10, mild disability; 11-20, moderate disability; >20, severe disability)
Changes in migraine disability (HIT-6) | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with atogepant
  Changes in Headache Impact Test-6 questionnaire across treatment (continuous variable, 36-78 scale, higher scores indicates greater disability)
Changes in response to acute migraine treatment (m-TOQ) | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with atogepant
  Changes in migraine Treatment Optimization Questionnaire across treatment (continuous variable, 0-8 scale, higher score indicates higher acute therapy effectiveness)
Changes in allodynia (ASC-12) | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with atogepant
  Changes in Allodynia Symptoms Checklist-12 questionnaire across treatment (continuous variable, 0-24 scale, higher score indicates more severe allodynia)
Changes in quality of life across atogepant treatment (MSQ) | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with atogepant
  Changes in Migraine Specific Quality of life questionnaire across treatment (continuous variable, 0-100 scale, 100 indicates full functionality)
Changes in interictal burden across atogepant treatment (MIBS-4) | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with atogepant
  Changes in Migraine Interictal Burden Scale-4 questionnaire across treatment (continuous variable, 0-4 scale, 0 indicates no interictal burden, 1-2 mild level of interictal burden, 3 moderate interictal burden, 4 severe interictal burden)
Self-reported treatment effectiveness | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with atogepant
  Changes in Migraine Assessment of Current Therapy (Migraine-ACT) a 4-item questionnaire about treatment effectiveness and daily life repercussions, across treatment compared to baseline (continuous variable, 0-4 scale, higher scores indicates higher acute treatment effectiveness)
Percentage of patients with Medication overuse headache reverted during treatment | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with atogepant
  Percentage of patients with a baseline diagnosis of MOH reverted after 3 - 6 and 12 months of treatment (continuous variable)

OTHER OUTCOMES:
Changes in the number of monthly migraine days with aura (quantitative) | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with atogepant
  Changes in monthly migraine days with aura across treatment (continuous variable, through headache diary assessment)
Variation of duration of aura (qualitative) | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with atogepant
  Changes in duration of aura across atogepant treatment (continuous variable - minutes, assessed through headache diary)
Variation of type of aura (qualitative) | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with atogepant
  Changes in type of aura across atogepant treatment (qualitative variable - assessed through headache diary and anamnestic data collection)
MMDs reduction in patients Non-responders to mAbs | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with atogepant
  Change of monthly migraine days across treatment in those patients who did not respond to anti-CGRP mAbs (continuous variable)
Percentage of 50% Responders across treatment in patients Non-responders to mAbs | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with atogepant
  Percentage of 50% Responders across treatment in those patients who did not respond to anti-CGRP mAbs (continuous variable)
Menstrually-related migraine | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with atogepant
  Change in the number of menstrually-related attacks (according to ICHD-3) across treatment compared to baseline (continuous variable)
Change in self-reported effectiveness of treatment | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with atogepant
  Change in Patients Global Impression of Change (PGIC) questionnaire across treatment (continuous variable, scale 0-7, 1 very much improved, 2 much improved, 3 minimally improved, 4 no change, 5 minimally worse, 6 much worse, 7 very much worse)
Changes in migraine severity | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with atogepant
  Changes in migraine severity (continuous variable, 0-10 numerical rating scale, higher scores indicate higher severity)
Changes in migraine duration | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with atogepant
  Changes in migraine duration (continuous variable- hours- assessed through a paper diary)
Changes in duration of the most bothersome symptom(s) | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with atogepant
  Changes in duration of the most bothersome symptom(s) across treatment (continuous variable, minutes, assessed through a paper diary)
Changes in severity of the most bothersome symptom(s) | Baseline (T0) - 3 months (T3) - 6 months (T6) - 12 months (T12) of treatment with atogepant
  Changes in severity of the most bothersome symptom(s) across treatment (continuous variable: 0-10 scale, higher scores indicate higher severity )

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - SOD Centro Cefalee e Farmacologia Clinica, AOU Careggi, Florence
  - Fondazione Policlinico Campus Bio-Medico, Roma

REFERENCES:
- [Background] Pozo-Rosich P, Ailani J, Ashina M, Goadsby PJ, Lipton RB, Reuter U, Guo H, Schwefel B, Lu K, Boinpally R, Miceli R, De Abreu Ferreira R, McCusker E, Yu SY, Severt L, Finnegan M, Trugman JM. Atogepant for the preventive treatment of chronic migraine (PROGRESS): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2023 Sep 2;402(10404):775-785. doi: 10.1016/S0140-6736(23)01049-8. Epub 2023 Jul 26. PMID 37516125
- [Background] Goadsby PJ, Dodick DW, Ailani J, Trugman JM, Finnegan M, Lu K, Szegedi A. Safety, tolerability, and efficacy of orally administered atogepant for the prevention of episodic migraine in adults: a double-blind, randomised phase 2b/3 trial. Lancet Neurol. 2020 Sep;19(9):727-737. doi: 10.1016/S1474-4422(20)30234-9. PMID 32822633
- [Background] Schwedt TJ, Lipton RB, Ailani J, Silberstein SD, Tassorelli C, Guo H, Lu K, Dabruzzo B, Miceli R, Severt L, Finnegan M, Trugman JM. Time course of efficacy of atogepant for the preventive treatment of migraine: Results from the randomized, double-blind ADVANCE trial. Cephalalgia. 2022 Jan;42(1):3-11. doi: 10.1177/03331024211042385. Epub 2021 Sep 14. PMID 34521260
- [Background] Tassorelli C, Nagy K, Pozo-Rosich P, Lanteri-Minet M, Sacco S, Nezadal T, Guo H, De Abreu Ferreira R, Forero G, Trugman JM. Safety and efficacy of atogepant for the preventive treatment of episodic migraine in adults for whom conventional oral preventive treatments have failed (ELEVATE): a randomised, placebo-controlled, phase 3b trial. Lancet Neurol. 2024 Apr;23(4):382-392. doi: 10.1016/S1474-4422(24)00025-5. Epub 2024 Feb 13. PMID 38364831
- [Derived] Vernieri F, Iannone LF, Lo Castro F, Sebastianelli G, De Santis F, Corrado M, Marcosano M, Ornello R, Grazzi L, Montisano DA, De Cesaris F, Munafo A, Fofi L, Doretti A, Vaghi G, Pistoia F, Ferrandi D, Battistini S, Sacco S, Guerzoni S, Altamura C; Italian Headache Registry (RICe) Study Group. Effectiveness and tolerability of atogepant in the prevention of migraine: A real life, prospective, multicentric study (the STAR study). Cephalalgia. 2025 Apr;45(4):3331024251335927. doi: 10.1177/03331024251335927. Epub 2025 Apr 23. PMID 40267275